CLINICAL TRIAL: NCT06057389
Title: The Effects of Black Aronia Melanocarpa Extract Combined With a Energy-restricted Diet on Metabolic Indicators and Intestinal Microecology in Obese Individuals With Impaired Fasting Blood Glucose
Brief Title: The Effects of Aronia Melanocarpa Extract on Obese Individuals With Impaired Fasting Blood Glucose
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: I-23PJ329
Record Dates: First submitted 2023-09-14; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group: an energy-restricted diet + aronia melanocarpa extract
  Interventions: Dietary Supplement: aronia melanocarpa extract
- Control group (Placebo Comparator): control group: an energy-restricted diet + maltodextrin
  Interventions: Dietary Supplement: aronia melanocarpa extract

INTERVENTIONS:
Dietary Supplement: aronia melanocarpa extract — aronia melanocarpa extract (each capsule contains 150 mg of anthocyanins and 30 mg of flavonoidst；twice a day，one at a time) combined with an energy-restricted diet

SUMMARY:
Obesity is closely related to many chronic diseases such as hypertension, coronary heart disease, hyperlipidemia, type 2 diabetes, fatty liver, certain types of tumors, etc, which are associated with adverse health outcomes. Limiting energy intake is one of the most important treatment measures for weight loss. The fruits of Aronia melanocarpa (Aronia berries) have been found to show multiple bioactivities potentially beneficial to human health, including antidiabetic, anti-infective, antineoplastic, antiobesity, antioxidant and gut microbiota-regulating activities. Thus, it is worth investigating whether consumption of aronia melanocarpa extract have additional benefits in improving anthropometric indicators, glucose and lipid metabolism, inflammatory status, adipocyte cytokines, and intestinal microbiota in obese individuals on the basis of an energy-restricted diet.

Obese individuals will be divided into intervention group and control group in this 8-week trial. Both groups will be given an energy-restricted diet, with an additional dose of aronia melanocarpa extract in capsules in intervention group and an additional dose of maltodextrin in capsules in control group.

Fecal and blood samples from participants before and after the intervention will be collected for the analysis of gut microbiota, glucose and lipid metabolism, inflammatory status, and adipocyte cytokines

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40 years
* Simple obese individuals with stable body weight in the last three months before enrollment (28.0kg/m2 ≤ BMI <35.0kg/m2)
* Impaired fasting blood glucose: Within the last three months before enrollment, the venous fasting blood glucose was between 6.1 and 7.0 mmol/L, and the 2-hour postprandial blood glucose was<7.8 mmol/L and the glycated hemoglobin (HbA1c) was < 6.5%

Exclusion Criteria:

* Diagnosed patients with diabetes or those who use hypoglycemic drugs
* Patients with concomitant hyperthyroidism or hypothyroidism, or those taking thyroxine tablets
* Those who apply glucocorticoids within 12 weeks
* Individuals with suspected renal dysfunction (female: serum creatinine ≥ 84 µ mol/L; male: serum creatinine ≥ 104 µ mol/L) or suspected liver dysfunction (elevated transaminase >3 times normal or cirrhosis)
* Secondary obesity (such as thalamic diseases, pituitary diseases, Cushing's syndrome, etc.)
* Previous weight loss surgeries
* Pregnant or lactating individuals
* Individuals with confirmed mental illness or eating disorders
* Women with polycystic ovary syndrome
* Individuals who are allergic or intolerant to experimental products
* Lactose intolerant individuals
* Those who have taken probiotics and/or probiotic drugs or supplements within one month before enrollment
* Those who fail to use intervention agents according to the study protocol or have severely incomplete visit records

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-10-07 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
gut microbiota | 8 weeks
  High flux sequencing of fecal specimens
glucose metabolism | 8 weeks
  Fasting blood glucose (in mmol/L)
glucose metabolism | 8 weeks
  fasting insulin (in μIU/L)
glucose metabolism | 8 weeks
  glycosylated hemoglobin (in %)
lipid metabolism | 8 weeks
  total cholesterol (in mmol/L)
lipid metabolism | 8 weeks
  triglycerides (in mmol/L)
lipid metabolism | 8 weeks
  high-density lipoprotein cholesterol (in mmol/L)
lipid metabolism | 8 weeks
  low-density lipoprotein cholesterol (in mmol/L)
leptin | 8 weeks
  serum leptin (in ng/ml)
adiponectin | 8 weeks
  serum adiponectin (in μg/ml)
Inflammatory cytokine | 8 weeks
  serum interleukin-1 (in pg/mL)
Inflammatory cytokine | 8 weeks
  serum interleukin-6 (in ng/L)
Inflammatory cytokine | 8 weeks
  tumor necrosis factor-α (in pg/ml)
Inflammatory cytokine | 8 weeks
  hypersensitive C-reactive protein (in mg/L)

SECONDARY OUTCOMES:
Anthropometrics | 8 weeks
  Body weight (in kg)
Anthropometrics | 8 weeks
  waist circumference (in cm)
Anthropometrics | 8 weeks
  BMI in kg/m^2
body composition | 8 weeks
  including body fat (in %), fat-free mass (in kg)